CLINICAL TRIAL: NCT07176689
Title: A Single-Arm, Open-Label Phase 4 Study of Nirogacestat in Adult Premenopausal Females With Desmoid Tumors/Aggressive Fibromatosis (DT/AF)
Brief Title: Nirogacestat in Premenopausal Females With Desmoid Tumor/Aggressive Fibromatosis (DT/AF)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIR-DT-401; 2024-515215-21-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-31; First posted 2025-09-16 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-11

CONDITIONS: Desmoid Tumor; Aggressive Fibromatosis
Keywords: Nirogacestat; PF-03084014; GSI; gamma secretase inhibitor; notch pathway; Ogsiveo
MeSH Terms: conditions — Desmoid Tumors | interventions — nirogacestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nirogacestat (Experimental): Nirogacestat 150 mg by mouth, twice daily
  Interventions: Drug: Nirogacestat

INTERVENTIONS:
Drug: Nirogacestat — Nirogacestat oral tablet
  Other Names: PF-03084014; Ogsiveo

SUMMARY:
This study is being conducted to study how nirogacestat may affect the ovarian function of adult premenopausal women with progressing desmoid tumors/aggressive fibromatosis.

DETAILED DESCRIPTION:
Desmoid tumors, also referred to as aggressive fibromatosis, are rare, locally invasive, slow growing soft tissue tumors. Although considered benign because of their inability to metastasize, desmoid tumors can cause significant morbidity and occasionally mortality in patients.

Nirogacestat is a tumor inhibitor that works by slowing or stopping the growth of tumor cells. Nirogacestat is a tablet taken by mouth and has been approved in the USA for adult patients with progressing desmoid tumors who require systemic treatment.

This is an open-label study to characterize the incidence and ovarian function recovery rates of ovarian toxicity (OT) events and to evaluate the efficacy, safety, and tolerability of nirogacestat in postpubertal and premenopausal females with desmoid tumors (DT).

ELIGIBILITY:
Inclusion Criteria:

* Participant is female, postpubertal aged ≥18 and ≤40 years of age at the time of signing the informed consent and premenopausal at baseline. Premenopausal is defined as meeting all of the following: Estradiol >30 pg/mL. Follicle-stimulating hormone (FSH) <40 IU/L. Regular menses (e.g., menstrual cycle length of 21 to 35 days) for at least 3 menstrual cycles prior to signing informed consent
* Participant uses 1 highly effective non-hormonal contraceptive method, has a negative pregnancy test prior to first dose of study treatment), is not breastfeeding, agrees to not harvest or donate eggs for at least 90 days prior to and during the study
* Participant has histologically confirmed DT/AF with symptomatic or progressive disease requiring systemic treatment
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status ≤2 at screening
* Participant has adequate organ and bone marrow function.

Exclusion Criteria:

* Participant has known malabsorption syndrome or preexisting gastrointestinal conditions that may impair absorption of nirogacestat
* Participant has experienced any of the following within 6 months of signing informed consent: clinically significant cardiac disease (New York Heart Association Class III or IV), myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, or symptomatic pulmonary embolism.
* Participant has had lymphoma, leukemia, or any malignancy within the past 5 years at the time of informed consent, except for any locally recurring cancer that has been treated curatively (e.g., resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast), with no evidence of metastatic disease for 3 years at the time of informed consent.
* Participant has known hepatic impairment
* Participant previously received or is currently receiving gamma secretase inhibitors or anti-Notch antibody therapy
* Participant is currently using any treatment for DT/AF including tyrosine kinase inhibitors (TKIs) or any investigational treatment 28 days (or 5 half-lives, whichever is longer) prior to the first dose of study treatment
* Participant is currently using or anticipates using food or drugs that are known strong/moderate cytochrome P450 (CYP) 3A4 inhibitors, or strong CYP3A inducers within 14 days prior to the first dose of study treatment.
* Participant has a history of polycystic ovary syndrome, hypothalamic amenorrhea, severe endometriosis involving ovaries, family history of primary ovarian insufficiency, any chromosomal abnormality, mutation, gene variant or medical condition associated with early/premature menopause, including a history of OT while on a TKI
* Participant is currently using or has used hormonal contraception or ovarian suppression within 90 days prior to first dose of study treatment
* Participant has a history of heavy tobacco smoking (≥20 pack years) or is a current smoker (>1 pack per day)
* Participant has experienced other severe acute or chronic medical or psychiatric conditions within 1 year of signing informed consent.
* Participant is unable to comply with study related procedures (including, but not limited to, the completion of a menstrual diary and electronic patient-reported outcomes and ability to return to clinic for hormone level blood draws timed to the menstrual cycle (days 1-5)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2031-02-28 (Estimated); Study Completion 2031-03-30 (Estimated)

PRIMARY OUTCOMES:
Ovarian function recovery rate of ovarian toxicity (OT) treatment-emergent adverse events (TEAEs) | Up to 24 cycles (each cycle is 28 days) of treatment and up to 2 years in the Clinical Follow-up Period
  Ovarian function recovery is defined as achieving the resumption of ≥2 consecutive menstrual periods and an FSH level <30 mIU/mL with concomitant estradiol <80 pg/mL OR resumption of ≥2 consecutive menstrual periods and AMH level within normal range adjusted for age and pretreatment baseline OR a positive serum β-HCG pregnancy test.

SECONDARY OUTCOMES:
Incidence of OT TEAEs | Up to 24 cycles (each cycle is 28 days) of treatment and up to 2 years in the Clinical Follow-up Period
  OT is any new onset amenorrhea lasting ≥3 consecutive menstrual periods, FSH level ≥30 mIU/mL and a negative β-HCG pregnancy test.
Time to ovarian function recovery in participants with a TEAE of OT | Up to 24 cycles (each cycle is 28 days) of treatment and up to 2 years in the Clinical Follow-up Period
  Time to ovarian function recovery is evaluated in participants who had a TEAE of OT and is defined as the time it takes to resolve.
The incidence of adverse events (AEs) according to toxicities graded by National Cancer Institute (NCI) Common Technology Criteria for Adverse Events (CTCAE) Version 5 | Up to 24 cycles (each cycle is 28 days) of treatment and up to 2 years in the Clinical Follow-up Period

OTHER OUTCOMES:
Objective Response Rate (ORR) | First day of every 3 cycles (each cycle is 28 days) for up to 24 cycles of treatment and up to 1 year in the Clinical Follow-up Period
  Proportion of participants with Complete Response (CR) and Partial Response (PR) using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria
Duration of Response (DoR) for participants whose best response is CR or PR | First day of every 3 cycles (each cycle is 28 days) until disease progression is observed or death, whichever comes first, up to 24 cycles of treatment and up to 1 year in the Clinical Follow-up Period
  DoR is defined as the duration from the time of first assessment of CR or PR response (per RECIST v1.1) to the first date of disease progression or death (whichever comes first).
Disease Control Rate (DCR) for participants whose best response is CR, PR or Stable Disease (SD) | First day of every 3 cycles (each cycle is 28 days) for up to 24 cycles of treatment and up to 1 year in the Clinical Follow-up Period
  DCR is defined as the proportion of participants who have a best response of CR, PR, or SD.
Duration of Disease Control (DoDC) for participants whose best response is CR, PR or SD | First day of every 3 cycles (each cycle is 28 days) until disease progression is observed or death, whichever comes first, up to 24 cycles of treatment and up to 1 year in the Clinical Follow-up Period
  DoDC is defined as the duration from the start of study treatment until first date of disease progression or death (whichever comes first).
Progression Free Survival (PFS) | First day of every 3 cycles (each cycle is 28 days) until disease progression is observed or death, whichever comes first, up to 24 cycles of treatment and up to 1 year in the Clinical Follow-up Period
  PFS is defined at the start of study treatment until the date of assessment of progression or death by any cause. Progression will be determined radiographically using RESIST v1.1 performed by a local radiologist.
Changes in tumor volume from baseline assessed by MRI volumetric analysis performed locally | First day of every 3 cycles (each cycle is 28 days) up to 24 cycles and up to 1 year in the Clinical Follow-up Period
Change in T2 hyperintensity baseline assessed by MRI analysis performed locally | First day of every 3 cycles (each cycle is 28 days) up to 24 cycles and up to 1 year in the Clinical Follow-up Period
Characterization of serum nirogacestat concentrations assessed in sparse pharmacokinetic (PK) sampling (pre-dose and 1-hour post dose at Cycle 1 Day 1 only) and trough PK sampling (pre-dose at treatment period visits after Cycle 1 Day 1 | First day of every 3 cycles (each cycle is 28 days) up to 24 cycles of treatment
Pain severity using Brief Pain Index - Short Form (BPI-SF), question #3 | From 7 days prior to date of first dose of treatment through end of Cycle 2 (each cycle is 28 days), assessed up to 9 weeks
  BPI question #3 will measure worst pain in the last 24 hours using an 11-point numeric scale from 0 (no pain) to 10 (pain as bad as you can imagine)
Patient experience of desmoid tumors and nirogacestat | One interview will occur following treatment completion (on average approximately 2 years after study entry) and a second interview will occur at study completion (on average approximately 3 years after study entry)
  Two (2) optional 60-minute qualitative interviews using open-ended exploratory questions to elicit spontaneous responses will be transcribed and analyzed in an inductive/deductive method to identify themes in the data

CONTACTS AND LOCATIONS:
Overall Officials: Winette van der Graff, MD, Principal Investigator — The Netherlands Cancer Institute
Locations (19):
- Cliniques Universitaires Saint-Luc (CUSL), Brussels, Belgium
- Universitätsklinikum Mannheim, Mannheim Cancer Center, Mannheim, Germany
- Italy (5):
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" IRCCS IRST. S.r.l., Meldola, Forli-Cesena
  - Fondazione del Piemonte per l'Oncologia Istituto di Candiolo IRCCS, Candiolo, Torino
  - IRCCS Istituto Ortopedico Rizzoli, Bologna
  - Istituto Nazionale Tumori I.R.C.C.S- Fondazione G. Pascale, Napoli
  - Fondazione Policlinico Unversitario Campus Bio-Medico di Roma, Roma
- Netherlands (2):
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek Ziekenhuis (NKI-AVL), Amsterdam
  - LUMC, Leiden
- Spain (6):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario y Politecnico La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (4):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - University College London Hospitals NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
SpringWorks Therapeutics is committed to data transparency and sharing data to further research while maintaining the privacy and confidentiality of research participants. Pertinent patient-level data from completed registrational clinical trials will be made available by SpringWorks to qualified researchers upon approval of reasonable requests following de-identification/anonymization pursuant to applicable law.